CLINICAL TRIAL: NCT01435603
Title: Community Translation of a Lifestyle Intervention to Improve Health in Diabetes
Brief Title: Intervening in Diabetes With Healthy Eating, Activity, and Linkages To Healthcare - The I-D-HEALTH Study
Acronym: I-D-HEALTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Ronald Ackermann, Professor of Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STU00056501; R18DK083941 (NIH)
Record Dates: First submitted 2011-09-12; First posted 2011-09-16 (Estimated); Results first posted 2018-04-27 (Actual); Last update posted 2018-04-27 (Actual); Status verified 2016-10

CONDITIONS: Diabetes Mellitus; Hyperglycemia; Obesity; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Overnutrition; Nutrition Disorders; Overweight; Body Weight; Signs and Symptoms
Keywords: Prevention & Control; Hyperglycemia; Obesity; Diabetes Mellitus; Cost Benefit Analysis
MeSH Terms: conditions — Diabetes Mellitus; Hyperglycemia; Obesity; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Overnutrition; Nutrition Disorders; Overweight; Body Weight; Signs and Symptoms | interventions — Counseling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Lifestyle Advice (Active Comparator): Primary care-based identification of pre-diabetes and/or type 2 diabetes with standard clinical education (offered by participant's usual primary care providers) and brief lifestyle advice (delivered by a study Research Assistant).
  Interventions: Behavioral: Standard Lifestyle Advice
- Advice Plus Lifestyle Intervention (Experimental): Primary care-based identification of pre-diabetes and/or type 2 diabetes with standard clinical education (offered by participant's usual primary care providers) and brief lifestyle advice (delivered by a study Research Assistant) Plus access to an intensive group-based lifestyle intervention offered in a community setting.
  Interventions: Behavioral: Standard Lifestyle Advice; Behavioral: Advice Plus Lifestyle Intervention

INTERVENTIONS:
Behavioral: Standard Lifestyle Advice — Standard clinical education is offered routinely by the participant's usual primary care team. Primary care teams receive educational outreach visits and are provided with clinical recommendations for lifestyle and cardiovascular risk factor management. Brief lifestyle advice is delivered by a study Research Assistant at baseline, 6, 12, and 24 months.
  Other Names: Brief Lifestyle Advice
Behavioral: Advice Plus Lifestyle Intervention — Standard clinical education offered routinely by the participant's usual primary care team. Primary care teams receive educational outreach visits for lifestyle and cardiovascular risk factor management. Brief lifestyle advice delivered by a study research assistant at baseline, 6, 12, and 24 months. AND, participant offered free of charge access to an intensive lifestyle intervention offered in a community setting. Lifestyle interventions are delivered in community settings by lay instructors from community organizations who are centrally trained by the study team.
  Other Names: Plan Ahead Lifestyle Intervention; Intensive Lifestyle Intervention
  Arms: Advice Plus Lifestyle Intervention

SUMMARY:
The purpose of this study is to compare ways of giving advice and providing support to improve diet and physical activity in adult primary care patients with elevated body mass index and dysglycemia.

DETAILED DESCRIPTION:
This is a randomized comparative effectiveness trial to evaluate the health and economic effects of a community-based intensive lifestyle intervention for adult primary care patients with elevated body mass index and dysglycemia (either type 2 diabetes or pre-diabetes). The study will use qualitative and quantitative methods to assess reach, effectiveness, costs, adoption, implementation, and maintenance of a clinical-community partnership to offer intensive lifestyle intervention resources to eligible adult primary care patients.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older, AND
2. Body-mass index of ≥ 24 kg/m2, AND
3. Documented Dysglycemia: Either by verification of laboratory test (Fasting Plasma Glucose 100-125 mg/dl OR 2-hour Post-challenge Plasma Glucose 140-199 mg/dl OR A1c 5.7%-10.9%) OR confirmation of Type 2 diabetes mellitus by self-report with verification

Exclusion Criteria (any of the following):

Diseases/Conditions that could limit lifespan and/or increase risk with a lifestyle intervention:

1. Significant cardiovascular disease:

   * Uncontrolled hypertension: systolic blood pressure >180 mmHg or diastolic blood pressure >105 mmHg
   * A1c > 10.9%
   * Heart attack, stroke, or transient ischemic attack (TIA) in the past 6 months
   * Chest pain, dizziness, or fainting with physical exertion
2. Lung disease:

   * Chronic obstructive airways disease or asthma requiring home oxygen
3. Pregnancy
4. Any other known condition that could limit ability to become physically active or limit life span to <5 years

Exclusions related to metabolism:

1. Use of medications known to produce hyperglycemia
2. Known disease leading to abnormal glucose metabolism, other than diabetes mellitus, including Cushing's syndrome; acromegaly; pheochromocytoma; chronic pancreatitis

Exclusion for conditions or behaviors likely to affect the conduct of the study:

1. Unable or unwilling to provide informed consent
2. Unable to communicate with the pertinent research study staff
3. Unable to read written English or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2011-08; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald T. Ackermann, MD, MPH, Principal Investigator — Northwestern University (Illinois)
Locations (2):
- United States (2):
  - YMCA of Metro Chicago, Chicago, Illinois
  - McGaw YMCA, Evanston, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Liss DT, Finch EA, Gregory DL, Cooper A, Ackermann RT. Design and participant characteristics for a randomized effectiveness trial of an intensive lifestyle intervention to reduce cardiovascular risk in adults with type 2 diabetes: The I-D-HEALTH study. Contemp Clin Trials. 2016 Jan;46:114-121. doi: 10.1016/j.cct.2015.11.016. Epub 2015 Dec 2. PMID 26611433
- [Derived] Liss DT, Finch EA, Cooper A, Sheth A, Tejuosho AD, Lancki N, Ackermann RT. One-year effects of a group-based lifestyle intervention in adults with type 2 diabetes: A randomized encouragement trial. Diabetes Res Clin Pract. 2018 Jun;140:36-44. doi: 10.1016/j.diabres.2018.03.030. Epub 2018 Mar 27. PMID 29596950

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Potential participants were prescreened on the phone and attended a baseline visit for further screening and enrollment.
Groups:
- Standard Lifestyle Advice: Primary care-based identification of pre-diabetes and/or type 2 diabetes with standard clinical education (offered by participant's usual primary care providers) and brief lifestyle advice (delivered by a study Research Assistant).
  Standard Lifestyle Advice: Standard clinical education is offered routinely by the participant's usual primary care team. Brief lifestyle advice is delivered by a study Research Assistant at baseline, 6, 12, and 24 months.
- Advice Plus Lifestyle Intervention: Primary care-based identification of pre-diabetes and/or type 2 diabetes with standard clinical education (offered by participant's usual primary care providers) and brief lifestyle advice (delivered by a study Research Assistant) Plus access to an intensive group-based lifestyle intervention offered in a community setting.
  Standard Lifestyle Advice: See "Standard Lifestyle Advice" arm.
  Advice Plus Lifestyle Intervention: Standard clinical education offered by the participant's usual primary care team. Brief lifestyle advice delivered by a study research assistant at baseline, 6, 12, and 24 months. AND, participant offered free of charge access to an intensive lifestyle intervention offered in a community setting. Lifestyle interventions are delivered in community settings by lay instructors from community organizations who are centrally trained by the study team.
Period: Overall Study
Arm/Group | Standard Lifestyle Advice | Advice Plus Lifestyle Intervention
Started | 167 | 164
Completed | 128 | 129
Not Completed | 39 | 35

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Lifestyle Advice | Advice Plus Lifestyle Intervention | Total
Number analyzed (Participants) | 167 | 164 | 331
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 124 | 125 | 249
  >=65 years | 43 | 39 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (12.2) | 57.1 (10.6) | 56.9 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 85 | 166
  Male | 86 | 79 | 165
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 43 | 48 | 91
  Not Hispanic or Latino | 124 | 116 | 240
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 9 | 6 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 54 | 50 | 104
  White | 63 | 62 | 125
  More than one race | 4 | 2 | 6
  Unknown or Not Reported | 37 | 44 | 81
Region of Enrollment [Number; unit: participants]
  United States | 167 | 164 | 331

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Body Weight
Description: (Body weight at 12 months subtracted from baseline body weight) divided by baseline body weight. Negative numbers indicate a weight loss.
Time Frame: Baseline to 12 months
Population: Participants who completed weight measurements at the baseline and 12 month exam
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Standard Lifestyle Advice | Advice Plus Lifestyle Intervention
Number analyzed (Participants) | 128 | 129
percentage of change | -0.15 (4.05) | -1.42 (4.45)
Statistical Analysis 1: Comparison: Standard Lifestyle Advice vs Advice Plus Lifestyle Intervention; Test type: Superiority; p = 0.017, Regression, Linear; Slope = -1.273

2. Secondary Outcome: Incremental Costs
Description: The study will capture direct medical, direct non-medical, and indirect costs from individual participants. Mean changes in these costs will be compared across randomized study arms.
Time Frame: 6, 12, and 24 months
Reporting Status: Not Posted

3. Secondary Outcome: Changes in Health State Utility
Description: The study collects individual participant survey data that will include the Medical Outcomes Study Short Form-12 health-related quality of life questionnaire. Responses from the questionnaire are used to construct a validated numerical score that expresses global health-related quality of life across a range of 0 (death) to 1 (perfect health). Changes in this indicator will be evaluated.
Time Frame: Baseline to 6,12, and 24 months
Reporting Status: Not Posted

4. Secondary Outcome: Percent Change in Body Weight
Time Frame: Baseline to 6 and 24 months
Reporting Status: Not Posted

5. Secondary Outcome: Percent Change in Blood Total Cholesterol
Time Frame: Baseline to 6, 12, and 24 months
Reporting Status: Not Posted

6. Secondary Outcome: Percent Change in A1c
Time Frame: Baseline to 6, 12, and 24 months
Reporting Status: Not Posted

7. Secondary Outcome: Percent Change in Blood Pressure
Time Frame: Baseline to 6, 12, and 24 months
Reporting Status: Not Posted

8. Secondary Outcome: Percent Change in Dietary Composition
Time Frame: Baseline to 6, 12, and 24 months
Reporting Status: Not Posted

9. Secondary Outcome: Percent Change in Physical Activity
Time Frame: Baseline to 6, 12, and 24 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Standard Lifestyle Advice | Advice Plus Lifestyle Intervention
All-Cause Mortality (participants affected / at risk) | 1/167 | 0/164
Serious Adverse Events (participants affected / at risk) | 10/167 | 10/164
Other Adverse Events (participants affected / at risk) | 0/167 | 0/164
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Lifestyle Advice (N=167) | Advice Plus Lifestyle Intervention (N=164)
Hypoglycemia (severe: admitted to hospital, emergency room, or needed assistance by other person) (Endocrine disorders) | 4 | 4
Heart attack (myocardial infarction) (Cardiac disorders) | 1 | 1
Congestive Heart Failure (Cardiac disorders) | 1 | 1
Balloon angioplasty or Stenting of coronary arteries (Percutaneous transluminal coronary angioplasty (Surgical and medical procedures) | 2 | 3
Stroke (transient ischemic attack, cerebral ischemia/hemorrhage, or cerebrovascular accident) (Nervous system disorders) | 1 | 1
Cardiac Arryhythmia (atrial fibrillation or flutter) (Cardiac disorders) | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 3 | 2

LIMITATIONS AND CAVEATS:
Over the 1 year measurement period, we experienced significant loss to follow-up in this diverse, predominantly low-income sample. We were only able to measure the primary outcome, body weight, on 257 of 331 participants at the 12 month visit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No